CLINICAL TRIAL: NCT06088316
Title: Efficacy of Amoxicillin-Esomeprazole High Dose Dual Therapy Compared to Levofloxacin Containing Triple Therapy for the Eradication of Helicobacter Pylori in a Tertiary Care Hospital: A Single-blind Randomized Controlled Trial
Brief Title: Efficacy of Amoxicillin-Esomeprazole HDDT Compared to Levofloxacin Triple Therapy for H. Pylori Eradication: A RCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Salman Rafat, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4270
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Helicobacter Pylori Infection; Helicobacter Pylori Eradication
Keywords: Helicobacter pylori; Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Intervention Model Description: participants will be randomly assigned into two groups- Group A & Group B. Group A will receive amoxicillin-esomeprazole high dose dual therapy for 14 days.
  Group B will receive levofloxacin containing triple therapy for 14 days. dyspeptic symptoms,drug side effects & H.pylori eradication rates will be compared between two groups.
Who Masked: Participant
Masking Description: Participants will be unaware about which group of treatment they are getting but the investigator will know about the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group-A (Experimental): Group A will receive amoxicillin-esomeprazole high dose dual therapy that is amoxicillin 1gm 8 hourly after meal & esomeprazole 40mg 8 hourly 30 minutes before meal for 14 days.
  Interventions: Drug: group A : Amoxicillin Esomeprazole HDDT
- Group-B (Active Comparator): Group-B patients will receive levofloxacin containing triple therapy that is Levofloxacin 500mg once daily after meal, Amoxicillin 1gm 12 hourly after meal & Esomeprazole 20mg 12 hourly 30 minutes before meal for 14 days.
  Interventions: Drug: group-B : Levofloxacin triple therapy

INTERVENTIONS:
Drug: group A : Amoxicillin Esomeprazole HDDT — Group A - Amoxicillin 1gm 8 hourly after meal & esomeprazole 40mg 8 hourly 30 minutes before meal for 14 days.
  Group-B - Levofloxacin 500mg once daily after meal, Amoxicillin 1gm 12 hourly after meal & Esomeprazole 20mg 12 hourly 30 minutes before meal for 14 days.
  Arms: Group-A
Drug: group-B : Levofloxacin triple therapy — Group-B - Levofloxacin 500mg once daily after meal, Amoxicillin 1gm 12 hourly after meal & Esomeprazole 20mg 12 hourly 30 minutes before meal for 14 days.
  Arms: Group-B

SUMMARY:
The goal of this clinical trial is to compare the efficacy of two different therapeutic regimen for the treatment of Helicobacter pylori infected dyspeptic patients. The aim is -

1. To identify the percentage of H. pylori infection among dyspeptic patients
2. To compare the efficacy of amoxicillin-esomeprazole high dose dual therapy with levofloxacin containing triple therapy for the eradication of Helicobacter pylori.

Participants will be screened on the basis of two different test (stool antigen test & endoscopy with rapid urease test) to detect H. pylori infection. Who are positive on both tests will be finally enrolled in the study and randomized into two groups . one group will receive amoxicillin & esomeprazole for 14 days in higher dose. The other group will receive amoxicillin, levofloxacin & esomeprazole for 14 days in usual dose.

Dyspeptic symptoms will be recorded before & after treatment. Side effects of drugs will also be recorded. Finally 1 month after completion of treatment , H.pylori status will be cheeked by stool antigen test and results will be compared between two groups.

DETAILED DESCRIPTION:
Introduction:

Helicobacter pylori infection is one of the most common infections worldwide and represents a major cause of gastritis, gastric and duodenal ulcers, mucosa-associated lymphoid tissue lymphoma. Moreover, H. pylori is recognized as a class 1 carcinogen by the International Agency for Research on cancer & WHO. It is the most important risk factor for developing gastric cancer, the timely elimination of which could lead to a 75% reduction in risk.

H. pylori infection higher in developing countries as compared to industrially developed countries and the prevalence varies between populations and between groups within the same population.According to a recent meta-analysis Bangladesh has the highest prevalence of H. pylori infection among Asian countries,86%

H. pylori antimicrobial resistance is an urgent, global issue. In addition to clarithromycin, resistance to metronidazole and fluoroquinolones has also increased worldwide . A recent study in Bangladesh showed clarithromycin, metronidazole & levofloxacin resistance at 39.3% ,94.6% and 66.1% respectively. On the contrary, amoxicillin resistance is quite low, 3.6%.

Since its discovery, various H. pylori eradication regimens have been investigated around the world with variable efficacy. Recent Maastricht's VI guideline recommends susceptibility testing before prescribing 1st line treatment if possible. Otherwise, bismuth or non-bismuth quadruple therapy followed by levofloxacin containing triple or quadruple therapy for 14 day is recommended for the treatment of H. pylori. Although these treatment regimens provide acceptable H. pylori eradication rates, dual & triple resistance to antibiotics adversely affects efficacy of these regimens. Moreover, these regimens can promote resistance, due to prolonged therapy with multiple antibiotics. A new strategy that can eradicate H. pylori as well as reduce the antibiotic exposure is required to prevent future antimicrobial resistance.

Amoxicillin is a beta-lactam antibiotic that inhibits cell wall synthesis of actively replicating cells and acts in a time-dependent manner meaning the more time plasma amoxicillin level remains above MIC, better the efficacy. So increasing dosing frequency enhances the bactericidal action of amoxicillin. PPI reduces intra-gastric acidity. Increasing the dosing frequency of PPI maintains acid suppression effectively over 24hour period. This promotes H. pylori replication & facilitates amoxicillin action. High dose dual therapy with esomeprazole and amoxicillin could be an alternative for H. pylori eradication in an era of growing antimicrobial resistance.For this reason this study was designed to compare the efficacy of amoxicillin-esomeprazole high dose dual therapy with levofloxacin containing triple therapy for the eradication of H. pylori.

Research Question:

Is amoxicillin-esomeprazole high dose dual therapy non-inferior to levofloxacin containing triple therapy for eradication of Helicobacter pylori ?

General objective:

To compare the efficacy of amoxicillin-esomeprazole high dose dual therapy with levofloxacin containing triple therapy for the eradication of Helicobacter pylori in a tertiary care hospital.

Specific objectives:

1. To identify H. pylori infection on the basis of stool antigen test & rapid urease test among dyspeptic patients
2. To identify H. pylori status on the basis of stool antigen test 4 weeks after amoxicillin- esomeprazole high dose dual therapy.
3. To identify H. pylori status on the basis of stool antigen test 4 weeks after levofloxacin containing triple therapy.
4. To assess the efficacy of amoxicillin-esomeprazole high dose dual therapy for H. pylori eradication
5. To assess the efficacy of levofloxacin containing triple therapy for H. pylori eradication
6. To compare the efficacy of amoxicillin-esomeprazole high dose dual therapy with levofloxacin containing triple therapy for H. pylori eradication

Study design: single-blind randomized controlled trial

Study population: Patients with dyspeptic symptoms attending the outpatient department of Gastroenterology, BSMMU-Dhaka meeting inclusion & exclusion criteria.

Inclusion criteria:

1. Age ≥ 18 years
2. Dyspeptic patients with positive Rapid urease test & stool antigen test
3. patients giving written informed consent

Exclusion criteria:

1. Treatment with proton pump inhibitor, H2-receptor antagonist, bismuth preparation within the last 2 weeks or antibiotics within 4 weeks prior to study.
2. Previous H. pylori eradication therapy
3. Complicated duodenal ulcer patients (active bleeding and perforation)
4. Patients with regular intake of NSAIDs or steroids.
5. Surgery that might affect gastric acid secretion (upper GI resection or vagotomy)
6. Known case of malignancy
7. Advanced Co-morbidities (e.g. CLD, CKD, cardio-respiratory failure, known thyroid disease)
8. participants who are pregnant, lactating or intend to become pregnant within the duration of the study.

Sample size calculation:

Numeric Results for Non-Inferiority Tests for the Ratio of Two Proportions Test Statistics: Ferrington & Manning Likelihood Score Test

Sample sizes of 32 in group 1 and 32 in group 2 achieve 81.041% power to detect a non-inferiority margin ratio in the group proportions of 0.950. the reference group proportion is 0.8900. the treatment group proportion is assumed to be 0.8455 under the null hypothesis of inferiority. The power was computed for the case when the actual treatment group proportion is 1.0000. the test statistic used is the one-sided score test.The significance level of the test is 0.050.

Considering 10% dropout rate 35 samples will be collected in each group. Total sample size will be 70.

Data collection:

Consecutive Patients with dyspepsia diagnosed on the basis of relevant history will initially be enrolled in the study maintaining inclusion and exclusion criteria from the outpatient department of Gastroenterology, BSMMU. Fresh stool sample will be collected from all dyspeptic patients in sterile container for stool antigen test. Stool antigen test will be carried out by one step chromatographic immunoassay (CerTest Biotec S.L. spain). Positive patients of stool antigen test will further undergo endoscopy of upper GIT after proper evaluation & ensuring that the patient is fit for endoscopy. Endoscopy will be performed by an experienced senior consultant & assisted by researcher himself using Olympus GIF-H190 endoscopy machine. Any mucosal lesion (e.g. gastritis, gastric ulcer, duodenal ulcer, erosion) will be noted in data sheet & biopsy (one from the antrum & one from corpus) will be taken for rapid urease test. Additional biopsy will also be taken for suspicious looking lesion. Rapid urease test will be carried out by RUT media obtained from department of microbiology. It will be composed of 40% urea solution, 0.01% neutral red and distilled water.it will be preserved at 37 degrees celsius in an incubator for 24 in the department of microbiology. The result will be considered positive when color change from yellow to pink. Patients who are positive on both SAT & RUT will be finally included in the study. Dyspeptic symptoms on a 5-point Likert scale will be recorded at enrolment.

Selected 70 patients will then randomly be assigned by computer generated method into two groups- Group A & Group B with 35 patients in each group.

Group A will receive amoxicillin-esomeprazole high dose dual therapy that is amoxicillin 1gm 8 hourly after meal & esomeprazole 40mg 8 hourly 30 minutes before meal for 14 days. Group-B patients will receive levofloxacin containing triple therapy that is Levofloxacin 500mg once daily after meal, Amoxicillin 1gm 12 hourly after meal & Esomeprazole 20mg 12 hourly 30 minutes before meal for 14 days.

Patients will be unaware about which group of treatment they are getting but the investigator will know about the treatment allocation.

Patients will be followed up at the end of therapy (day-14) for drug compliance (using drug compliance monitoring card and empty medicine strip) & for recording of any side effects either in person or over telephone. 1 month after completion of therapy, fresh stool sample will be collected from all patients for repeat stool antigen test & H. pylori eradication will be recorded for each group. Patients who had mucosal lesion at enrolment will also undergo repeat upper GI endoscopy for re-evaluation of mucosal lesion. Dyspeptic symptoms through 5point Likert score will be also recorded for each group 1 month after completion of therapy to cheek for any improvement or not.

Statistical analysis:

The following steps will be used to analyze the collected data:

* The entered data will be checked, verified and analyzed by IBM® SPSS® Statistics 25 (statistical program for social science) software.
* The data will be presented in tabular, figures and diagrammatical form.
* Appropriate statistical test will be applied for data analysis. Numeric data e.g. Age, Likert scale score for dyspepsia will be expressed as mean ± standard deviation and median (range) ,qualitative data e.g. sex, stool antigen test, endoscopy upper GIT will be expressed as frequency and percentage.
* Baseline characteristics of the study patients and outcomes will be evaluated using student's t-test, ANOVA, Chi-square test or Fisher's exact test, as appropriate. Factors influencing the efficacy of the eradication therapy were assessed by univariate & multivariate analysis
* A P-value less than 0.05 will be considered as significant at a 95% confidence interval (95% CI).

Quality assurance strategy This will be a single blinded randomized control trial. Extensive literature review will be done and investigator will be sufficiently trained. Inclusion and exclusion criteria will be strictly maintained. Every step of the study will be carried out under direct supervision of the guide. The completeness and quality of the collected data will be ensured by regular and routine supervision, checking and monitoring. Guide will randomly scrutinize the data collection procedure. Gathered information from patient will be checked and rechecked with medical record. Schedule meeting will be arranged with the guide and co-guide regularly to discuss the progress of data collection. Data cleaning will be done before editing in the computer for analysis. After obtaining results of one quarter of the study subjects, review meeting will be arranged with the guide and emerged issue will be addressed properly. Before entering data in computer for analysis random checking of 2% of data will be done by the guide. Irrelevant and inconsistent data will be discarded. After collection of data, meeting will be arranged with guide at weekly interval to discuss about the progress of thesis writing and submission.

Confidentiality:

All the information collected from the patients including the results of the laboratory tests will be kept as confidential under the responsibility of principal investigator. No one other than the investigators, regulatory authorities and institutional review board committee will have access to such information. Patient's identity will not be disclosed while analyzing or publishing the results of the study

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Dyspeptic patients with positive Rapid urease test & stool antigen test
3. patients giving written informed consent

Exclusion Criteria:

1. Treatment with proton pump inhibitor, H2-receptor antagonist, bismuth preparation within the last 2 weeks or antibiotics within 4 weeks prior to study.
2. Previous H. pylori eradication therapy
3. Complicated duodenal ulcer patients (active bleeding and perforation)
4. Patients with regular intake of NSAIDs or steroids.
5. Surgery that might affect gastric acid secretion (upper GI resection or vagotomy)
6. Known case of malignancy
7. Advanced Co-morbidities (e.g. CLD, CKD, cardio-respiratory failure, known thyroid disease)
8. participants who are pregnant, lactating or intend to become pregnant within the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy of amoxicillin-esomeprazole HDDT therapy with levofloxacin triple therapy for the eradication of Helicobacter pylori | 1 month after completion of eradication therapy
  Group A will receive amoxicillin-esomeprazole high dose dual therapy for 14 days. Group-B patients will receive levofloxacin containing triple therapy 14 days. 1 month after completion of therapy, fresh stool sample will be collected from all patients for repeat stool antigen test & H. pylori eradication will be recorded for each group. Eradication rate will be compared between two groups.

SECONDARY OUTCOMES:
Helicobacter pylori prevalence among dyspeptic patients | stool antigen test & rapid urease test will be done 14 days after stopping PPI ,H2 receptor antagonist,bismuth preparation
  To identify H. pylori infection on the basis of stool antigen test & rapid urease test among dyspeptic patients. patients tested positive on both tests will be considered H.pylori positive

OTHER OUTCOMES:
dyspeptic symptoms improvement in group A & group B | 1 month
  Dyspeptic symptoms through 5point Likert score will be recorded for each group at baseline & 1 month after completion of therapy to cheek for any improvement or not.
Endoscopic mucosal healing in group-A & group-B | 1 month
  Patients who had mucosal lesion at enrolment will undergo repeat upper GI endoscopy for re-evaluation of mucosal lesion 1 month after completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Salman Rafat, Mbbs, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu sheikh mujib medical university, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
All the collected IPD
Supporting Information: Study Protocol, ICF
Time Frame: starting 12 months after publication
Access Criteria: publishers ,any researcher interested in this field may have access